CLINICAL TRIAL: NCT03873623
Title: The TOGETHER Project - Transplant Organ Genomics to Help Prevent Rejection in Kidney Transplant Recipients With Realtime Assay Monitoring
Brief Title: The TOGETHER Project - Kidney
Acronym: TOGETHER
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark Stegall, Principal Investigator, Mayo Clinic
Other Study IDs: 16-003159
Record Dates: First submitted 2019-03-12; First posted 2019-03-13 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Kidney Transplant Rejection
Keywords: Kidney transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 7.5 ml of blood assays will be collected. Peripheral blood will be collected at 1, 4, 6, 9, and 12 months, as well as any for cause time points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney Transplant Recipients

SUMMARY:
Researchers are trying to develop a way to customize immunosuppression treatment, based on the results of a blood test that measures the risk of rejection.

ELIGIBILITY:
Inclusion Criteria:

* Conventional solitary kidney transplant (ABO compatible, crossmatch negative, not a kidney transplant simultaneously transplanted with another non-renal organ including heart, liver, lung or pancreas)
* Patients who have given informed consent and are willing to comply with the protocol, including the use of their specimens and data for subsequent research.

Exclusion Criteria:

* EBV -seronegative recipient
* ABO incompatible kidney transplants.
* Simultaneous kidney and extra-renal organ transplants including pancreas, liver, heart, lung, bone marrow transplantation, etc or prior recipient of non-renal transplant. Subjects who had previous extra renal transplants may be included in the study.
* Positive crossmatch kidney transplants (T cell crossmatch >100, B flow cytometric crossmatch >150).
* Participating in other clinical trials
* Any kidney transplant recipient < 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
To correlate the findings of TruGraf (a peripheral blood RNA signature that has been shown to correlate with rejection in renal allografts) with rejection episodes in renal transplant patients . | 3 years
  The study will validate the ability of a peripheral blood assay to assess the risk of rejection and determine the role this assay will have in immunosuppression monitoring in our patients at Mayo Clinic (3 sites).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stegall, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials